CLINICAL TRIAL: NCT04887129
Title: COV-IDD: Testing for COVID-19 in High Risk Children With Intellectual and Developmental Disabilities
Brief Title: Testing for COVID-19 in High Risk Children With Intellectual and Developmental Disabilities (COV-IDD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Foxe, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00005294; OT2HD107553-01 (NIH)
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students and staff at Mary Cariola Center (Experimental): All students enrolled at the Mary Cariola Center in Rochester, NY. All staff working at the Mary Cariola Center in Rochester, NY.
  Interventions: Diagnostic Test: COVID-19 RT-PCR test; Other: COVID-19 Vaccine Education Campaign

INTERVENTIONS:
Diagnostic Test: COVID-19 RT-PCR test — Participating individuals (students and employees) will be tested for COVID-19 (RT-PCR) using a specimen collected using a mid-turbinate swab.
  This asymptomatic testing regime starts on or after (if scheduling testing requires this to begin on a different day) enrollment and is repeated every 5-14 days for up to 16 months . Anyone testing positive is followed up as described below for symptomatic individuals.
  Those presenting with symptoms will be also tested for COVID-19 (RT-PCR). Those with negative test results will return to the asymptomatic testing protocol.
  Students who test positive are retested then 3 days until two negative tests. Employees who test positive also be tested every 3 days until two negative tests.
Other: COVID-19 Vaccine Education Campaign — Utilizing information from focus groups, the investigators will develop and deploy an educational campaign aimed at improving vaccine hesitancy and student health

SUMMARY:
The purpose of this study is to understand how to prevent COVID-19 spread in a school like the Mary Cariola Center (MCC) in Rochester, NY by answering questions like these: how do activities in the school alter chances of infection? Are there people infected with the COVID-19 virus who have no symptoms? How is spread of COVID-19 affected by vaccination rates? Is there any hesitancy to get the vaccine and what are the reasons? This information will be used to help keep the school open and the students and staff safe.

Eligible participants are those that work at the Mary Cariola Center (MCC) and interact with the students at MCC who have a high risk of infection from COVID-19.

The study lasts for up to 16 months.

ELIGIBILITY:
Inclusion Criteria:

Students:

* IDD Student of the Mary Cariola Center
* Age 3 - 18
* Have a parent/guardian who can give informed consent
* In the judgement of the Mary Cariola Medical Staff will be able to safely participate in the study procedures (nasal swab, phlebotomy)

Staff

* Age 18 - 72
* Able give informed consent
* Anticipated duration of remaining employment less than 1 month (e.g. retiring)
* Must be willing to participate in RT-PCR and antibody testing

Exclusion Criteria:

Students

* Contraindication to nasal swab
* Contraindication to phlebotomy (e.g. anticoagulated, bleeding diathesis)

Staff

* Contraindication to nasal swab
* Contraindication to phlebotomy (e.g. anticoagulated, bleeding diathesis)

Ages: 3 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Cariola Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Students; Staff: All students enrolled at the Mary Cariola Center in Rochester, NY. All staff working at the Mary Cariola Center in Rochester, NY.
Period: Overall Study
Arm/Group | Students | Staff
Started | 59 (of the 392 participants who started the study, 332 were staff and 59 were students.) | 333
Completed | 48 (Of the participants who completed the study, 243 were staff and 48 were students. 24 staff and 0 students were lost to follow-up. 57 staff and 9 students were withdrawal by subject. 9 staff and 2 students were unknown.) | 243
Not Completed | 11 | 90
Not completed — Lost to Follow-up | 0 | 24
Not completed — Withdrawal by Subject | 9 | 57
Not completed — Other | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Students | Staff | Total
Number analyzed (Participants) | 59 | 333 | 392
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [6 to 15] | 33 [27 to 43] | NA [NA to NA] — The two arms reported here are students and staff, children and adults, respectively. Therefore, it is not meaningful to combine the age data and calculate a median for the all participants.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data was missing for 14 students and 44 staff.
  Participants
    number analyzed (Participants) | 45 | 289 | 334
    Female | 14 | 253 | 267
    Male | 31 | 36 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 14 | 17
  Not Hispanic or Latino | 41 | 274 | 315
  Unknown or Not Reported | 15 | 45 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 8 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 38 | 46
  White | 32 | 225 | 257
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 14 | 52 | 66
Region of Enrollment [Number; unit: participants]
  United States | 59 | 333 | 392

OUTCOME MEASURES:

1. Primary Outcome: Number Infected With COVID-19
Description: Number of students or staff who test positive for COVID-19 at least once using a nasal swab test.
Time Frame: 16 months
Population: 12 staff members did not have a valid test for COVID
Measure: Count of Participants; unit: Participants
Groups:
- Students; Staff: All students enrolled at the Mary Cariola Center in Rochester, NY.
Arm/Group | Students | Staff
Number analyzed (Participants) | 59 | 321
Participants | 29 | 141

2. Primary Outcome: Change in the Percentage of Participants Reporting Anxiety
Description: Anxiety will be measured using the PROMIS-29 assessment. Participants were classified within normal range, mild, moderate or severe. They were counted as having anxiety if they were moderate or severe.
Time Frame: baseline to 16 months
Population: 29 students did not have data collected at 16 months. 165 adults did not have data collected at 16 months.
Measure: Number; unit: percentage of participants
Groups:
- Staff: All staff working at the Mary Cariola Center in Rochester, NY.
Arm/Group | Students | Staff
Number analyzed (Participants) | 30 | 168
percentage of participants | 11.7 | -0.7

3. Primary Outcome: Change in the Percentage of Participants Classified as Depressed
Description: Depression was measured using the PROMIS-29 assessment. Students or staff were classified within normal range, mild, moderate or severe. They were counted as having depression if they were moderate or severe.
Time Frame: baseline to 16 months
Population: 29 students did not have data collected at 16 months. 165 adults did not have data collected at 16 months.
Measure: Number; unit: percentage of participants
Arm/Group | Students | Staff
Number analyzed (Participants) | 30 | 168
percentage of participants | -0.8 | 3.5

4. Primary Outcome: Change in the Percentage of Participants Classified With Fatigue
Description: Fatigue will be measured using the PROMIS-29 assessment. Participants were classified within normal range, mild, moderate or severe. They were counted as having fatigue if they were moderate or severe.
Time Frame: baseline to 16 months
Population: 29 students did not have data collected at 16 months. 165 adults did not have data collected at 16 months.
Measure: Number; unit: percentage of participants
Arm/Group | Students | Staff
Number analyzed (Participants) | 30 | 168
percentage of participants | 2.3 | 11.8

5. Primary Outcome: Change in Percentage of Participants With Deficits in Social Functioning
Description: Social functioning will be measured using the PROMIS-29 assessment. Participants were classified within normal range, mild, moderate or severe. They were counted as having social functioning deficits if they were moderate or severe.
Time Frame: baseline to 16 months
Population: 29 students did not have data collected at 16 months. 165 adults did not have data collected at 16 months.
Measure: Number; unit: percentage of participants
Arm/Group | Students | Staff
Number analyzed (Participants) | 30 | 168
percentage of participants | 1.7 | 1.2

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Students | Staff
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/333
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/333
Other Adverse Events (participants affected / at risk) | 0/59 | 5/333
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Students (N=59) | Staff (N=333)
faintness (General disorders) | 0 | 1
Bite (Injury, poisoning and procedural complications) | 0 | 1
false positive COVID test (Infections and infestations) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04887129/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT04887129/SAP_001.pdf
  • Informed Consent Form (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT04887129/ICF_002.pdf